CLINICAL TRIAL: NCT03145194
Title: A Randomised Mechanistic Study Comparing the Effects of Different Anti-platelet Combinations (Ticagrelor vs. Placebo/ Clopidogrel) With Aspirin in Patients Presenting With Anterior STEMI Treated With Primary PCI
Brief Title: TIMES: Ticagrelor vs. Placebo/ Clopidogrel With Aspirin in Anterior STEMI Patients Treated With Primary PCI
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Papworth Hospital NHS Foundation Trust (Other Government)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: P01910
Record Dates: First submitted 2017-04-13; First posted 2017-05-09 (Actual); Last update posted 2017-05-30 (Actual); Status verified 2017-05

CONDITIONS: ST Elevation Myocardial Infarction
MeSH Terms: conditions — ST Elevation Myocardial Infarction | interventions — Ticagrelor

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Double blind until the point of primary endpoint.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ticagrelor (Experimental): Patients will receive Ticagrelor 180mg (2 x 90mg tablets)
  Interventions: Drug: Ticagrelor
- Placebo (Placebo Comparator): Patients will receive Placebo (2 matching tablets)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Ticagrelor — 2 x 90mg Ticagrelor tablets
  Arms: Ticagrelor
Other: Placebo — 2 x matching placebo tablets
  Arms: Placebo

SUMMARY:
This is a single-centred, double blind randomized controlled trial comparing ticagrelor with placebo in clopidogrel and aspirin loaded patients.

DETAILED DESCRIPTION:
The very early benefit of ticagrelor in STEMI is co-mediated by adenosine cardioprotection maintaining/ improving myocardial microcirculatory function, as well as via platelet inhibition or possibly other pleiotropic effects.

Ticagrelor increases circulating adenosine by reducing cellular re-uptake. Adenosine is a cardioprotective agent that utilizes cellular survival kinase pathways that may have beneficial effects on the microcirculation and myocardium in patients presenting with STEMI. Adenosine is currently used as a treatment for no-reflow and improves MVO post-STEMI when administered during PPCI. A recent study of healthy volunteers has confirmed that non-invasive coronary flow is augmented by ticagrelor and that this is mediated by adenosine. The Investigators propose that the very early beneficial effects of Ticagrelor in ACS may be adenosine mediated cardioprotection, rather than only due to an antiplatelet effect. This important research is original and a natural progression of the ticagrelor story. It expands the adenosine hypothesis and mode of action of ticagrelor and addresses a novel cardioprotective/ microcirculatory mechanism of action.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of informed verbal consent prior to any study specific procedures taking place with written consent confirmed prior to in-patient cardiac MRI.
2. Male or female adult patient aged 18 - 90 years old
3. Anterior STEMI (ST elevation ≥ 2mmHg in contiguous chest leads) with chest pain symptom onset < 12 hours

Exclusion Criteria:

1. Cardiogenic shock*
2. Previous anterior myocardial infarction
3. Unfavourable coronary anatomy for PCI: left main / surgical or distal coronary disease
4. Already prescribed Ticagrelor at the time of admission
5. Factors affecting study drug administration/ absorption: vomiting or allergy
6. Concomitant use of potent CYP3A4 inhibitors/ inducers (e.g ketoconazole and rifampicin) or CYP3A4 substrates with a narrow therapeutic window (e.g. cisapride and ergot alkaloids) or simvastatin / lovostatin >40mg oral dose.
7. Severe bleeding diathesis or current active bleeding*
8. History of intracranial haemorrhage
9. Moderate or Severe hepatic impairment
10. Severe asthma or bradycardia/ complete heart block (contraindications to adenosine)*
11. Severe co-morbidity with a life expectancy < 3 months.
12. Women of child bearing potential (as determined by direct questioning of the patient to confirm and this will be documented in the medical notes).

    * Patients that are found to have any excluding factor (e.g., unfavourable coronary anatomy for PCI) or develop any excluding factor (e.g., vomiting or cardiogenic shock) before the point of final IMR assessment will be discontinued from the study and followed up at discharge and by telephone at 3 and 12 months for adverse event monitoring purposes only.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2017-01-30 (Actual); Primary Completion 2018-11-30 (Estimated); Study Completion 2019-11-30 (Estimated)

PRIMARY OUTCOMES:
Index of Myocardial Resistance (IMR) | Baseline to end of PPCI procedure.
  To compare final Index of Myocardial Resistance (IMR) at the end of the PPCI procedure between the two arms.

SECONDARY OUTCOMES:
Baseline IMR and change in IMR during PPCI | Baseline to end of PPCI procedure.
  To compare between the two arms.
ACF and AMR pre/post PPCI | Baseline to end of PPCI procedure.
  To compare between the two arms.
TIMI flow and TMBG pre/post PPCI | Baseline to end of PPCI procedure.
  To compare between the two arms.
ST segment resolution | Baseline to end of PPCI procedure.
  To compare between the two arms.
OCT quantified clot volume pre/post PPCI | Baseline to end of PPCI procedure.
  To compare between the two arms.
Cardiac troponin - I and CKMB levels at 0, 12 and 24 hours | Baseline to 24 hours.
  To compare between the two arms.
Cardiac MRI microvascular obstruction between 24-48 hours and infarct size at 3 months | Baseline to 3 months.
  To compare between the two arms.

OTHER OUTCOMES:
Creatinine levels (eGRF) at 0, 12 and 24 hours | Baseline to 24 hours.
  Safety endpoint.
NYHA Functional Classification and CCS Angina Grading Scale | Discharge to 12 months.
  Clinical grading scales of heart failure and angina.
Plasma Ticagrelor levels at the point of final IMR measurement and in-patient Cardiac MRI. | End of PPCI procedure to 24-48 hours.
  This will explore if the IMR differences observed are related to individual differences in drug levels.
Plasma Adenosine levels at the point of final IMR measurement and in-patient Cardiac MRI | End of PPCI procedure to 24-48 hours.
  This will explore if the IMR differences observed are related to individual differences in adenosine levels.
Multiplatelet® ADP aggregation assessment of platelet reactivity at the point of final IMR measurement and in-patient Cardiac MRI | End of PPCI procedure to 24-48 hours.
  This will explore if the IMR differences observed are related to individual differences in platelet reactivity levels.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Hoole, Principal Investigator — Papworth Hospital NHS Foundation Trust
Locations (1):
- Papworth Hospital NHS Foundation Trust, Papworth Everard, Cambridge, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Aetesam-Ur-Rahman M, Brown AJ, Jaworski C, Giblett JP, Zhao TX, Braganza DM, Clarke SC, Agrawal BSK, Bennett MR, West NEJ, Hoole SP. Adenosine-Induced Coronary Steal Is Observed in Patients Presenting With ST-Segment-Elevation Myocardial Infarction. J Am Heart Assoc. 2021 Jul 6;10(13):e019899. doi: 10.1161/JAHA.120.019899. Epub 2021 Jun 30. PMID 34187187